CLINICAL TRIAL: NCT06644105
Title: Pharmacokinetic Study of Cefditoren Pivoxil in Breast Milk and Blood of Lactating Women
Acronym: RID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West China Second University Hospital (Other)
Responsible Party: Principal Investigator, Yu Qin, Principal Investigator, West China Second University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2024004-TBTLPZ
Record Dates: First submitted 2024-10-11; First posted 2024-10-16 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Medication Safety; Drug Safety; Drug Metabolism
MeSH Terms: interventions — cefditoren pivoxil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- subjects took cefditoren pivoxil tablets 200mg after a meal (Experimental): take cefditoren pivoxil tablets 200mg after a meal
  Interventions: Drug: cefditoren pivoxil tablets

INTERVENTIONS:
Drug: cefditoren pivoxil tablets — took cefditoren pivoxil tablets 200mg after

SUMMARY:
The goal of this clinical trial is to provide a theoretical basis for the rational use of cefditoren pivoxil in lactating women by conducting a pharmacokinetic study of cefditoren in the blood and milk of these women. The main questions it aims to answer are:

Can lactating women use cefditoren pivoxil? Is cefditoren distributed in breast milk?

12 Participants will:

Take cefditoren pivoxil tablets 200mg after a meal, and collect breast milk and plasma over certain time periods.

DETAILED DESCRIPTION:
This study is a single-center, single-sequence, open-label pharmacokinetic study involving Chinese healthy lactating subjects. It aims to investigate the exposure of cefditoren in blood and milk in lactating women. The M/P (milk to plasma) ratio was estimated through the area under the plasma and milk concentration-time curves (AUC) [6], and the infant's exposure (Relative Infant Dose，RID) was estimated as the product of the actual milk production and the average milk drug concentration, normalized by body weight and expressed as a percentage of the mother's dose adjusted for body weight. By studying the pharmacokinetics of cefditoren in blood and milk, the study provides a theoretical basis for the rational use of cefditoren pivoxil in lactating women.

ELIGIBILITY:
Inclusion Criteria:

1. Lactating women, aged 25-45 years (inclusive) at the time of informed consent
2. Body Mass Index (BMI) of 19 to 28 kg/m^2 (inclusive)
3. weight not less than 45.0 kg
4. Physical examination results including vital signs (blood pressure, pulse, and body temperature), physical examination, laboratory tests (complete blood count, blood biochemistry, and urine routine), and 12-lead ECG are all normal or the abnormalities are not clinically significant
5. The subject has no plans for pregnancy or oocyte donation from the time of signing the informed consent until 3 months after the end of the trial, and is willing to take effective contraceptive measures
6. The subject is able to communicate well with the researcher and understands and is able to comply with the requirements of this study.

Exclusion Criteria:

1. Individuals found during screening to have clinically significant diseases (including but not limited to respiratory, circulatory, cardiovascular, digestive, hematological, endocrine, immune, skin, nervous system, carnitine deficiency, or congenital metabolic defects that can cause significant carnitine deficiency, and related diseases)
2. Those with a history of specific allergies (asthma, urticaria, eczema, etc.), or allergic constitution (such as those allergic to two or more drugs, foods), or known to be allergic to any component of cefditoren pivoxil tablets, especially the cephalosporin antibiotics and excipients
3. Acute diseases occurring from the screening period to before the study medication or concomitant medication use
4. Received surgical procedures (cesarean section excluded) within 3 months before screening, or planning to undergo surgical procedures during the study period
5. Abnormalities of clinical significance judged by a clinical physician based on comprehensive physical examination, ECG, vital signs, and laboratory tests (complete blood count, coagulation function, blood biochemistry, urine routine, pre-transfusion panel) during the screening period
6. Positive results in any of the tests for hepatitis B surface antigen (TP-trust), hepatitis C virus antibody, anti-human immunodeficiency virus antibody, or syphilis spirochete antibody
7. Use of any drugs that may interact with the test drug within 30 days before the first administration, including CYP3A4 inhibitors and inducers (such as inducers-barbiturates, carbamazepine, phenytoin, rifampicin, etc.
8. inhibitors-SSRI class antidepressants, cimetidine, cyclosporine, macrolides, verapamil, fluoroquinolones, pyrrolidine antifungal drugs, HIV protease inhibitors, etc.), CYP2C9 inhibitors and inducers (such as inhibitors-sulfamethoxazole, amiodarone, fluconazole, metronidazole, prednisone, etc.
9. inducers-apalutamide, darunavir, enzalutamide, letermovir, nevirapine, secobarbital, St. John's wort, etc.), antacids (such as omeprazole, rabeprazole, pantoprazole, ranitidine, famotidine, aluminum hydroxide, magnesium hydroxide, or sucralfate) and other drugs
10. Use of any prescription drugs, over-the-counter drugs, Chinese herbal medicine, or health products within 2 weeks before taking the study medication
11. Blood donation or significant blood loss (>400 mL), blood transfusion, or use of blood products within 3 months before screening
12. Received live or attenuated vaccines within 1 month before screening, or planning to receive live or attenuated vaccines during the trial period
13. Participated in any medical device clinical trials or drug clinical trials and used trial medical devices and/or drugs within 3 months before screening
14. Intolerant to venipuncture, fainting at the sight of blood or needles, or poor venous access for blood collection
15. Having special dietary requirements, lactose intolerance, inability to comply with the provided diet and corresponding regulations, or difficulty swallowing pills
16. Positive drug abuse screening, or a history of drug abuse within the past five years, or use of drugs within 3 months before screening, or positive urine drug screening results
17. Regular alcohol consumption within 3 months before screening, i.e., more than 2 units of alcohol per week (1 unit = 360 mL of beer with 5% alcohol content, or 45 mL of spirits with 40% alcohol content, or 150 mL of wine with 12% alcohol content), and/or unwilling to abstain from alcohol intake 48 hours before and during the hospital stay
18. An average daily smoking amount of more than 5 cigarettes within 3 months before screening, and/or unwilling to avoid the use of any tobacco products during the trial period
19. Consumption of any food or beverages rich in caffeine, poppy seeds and/or theophylline, theobromine, cocoa (such as coffee, strong tea, chocolate, and caffeinated carbonated beverages, cola, etc.) within 48 hours before taking the study medication, or consumption of any food or beverages rich in grapefruit (such as grapefruit juice) within 48 hours before taking the study medication, or engaging in vigorous exercise
20. Subjects who may not be able to complete the study for other reasons, or whom the researcher judges to have other reasons not suitable for participating in the trial.

Ages: 25 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2024-01-10 (Actual); Primary Completion 2024-01-24 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
the relative infant dose | within 12 hours after taking the medication
  estimated as the product of the actual milk production and the average milk drug concentration, normalized by body weight and expressed as a percentage of the mother's dose adjusted for body weight
the milk-to-plasma ratio | within 12 hours after taking the medication
  milk to plasma ratio

CONTACTS AND LOCATIONS:
Overall Officials: Qin yu, Principal Investigator — National Drug Clinical Trial Institution of West China Second Hospital
Locations (1):
- West China Second University Hospital, Chengdu, China

IPD SHARING:
Plan to Share IPD: Yes
The data that support the findings of this study are available from the corresponding author upon reasonable request.
Supporting Information: Study Protocol, ICF, CSR, Analytic Code